CLINICAL TRIAL: NCT04438200
Title: Niveles de Retinol Hepatico y óseo en cadáveres de Adolescentes y Adultos Guatemaltecos (Liver and Bone Retinol Levels in Guatemalan Adolescents and Adults)
Brief Title: Liver and Bone Retinol Levels in Guatemalan Adolescents and Adults
Acronym: GVAS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Newcastle University (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); HarvestPlus (Other); Institute of Nutrition of Central America and Panama (Other); INACIF (Unknown)
Responsible Party: Sponsor
Other Study IDs: VDACS-MF-0109-2019
Record Dates: First submitted 2020-03-23; First posted 2020-06-18 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-02

CONDITIONS: Vitamin A Deficiency; Vitamin A Toxicity; Hypervitaminosis A
Keywords: Retinol; Hypervitaminosis A; Hepatic Vitamin A; Guatemala
MeSH Terms: conditions — Vitamin A Deficiency; Hypervitaminosis A

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Liver Tissue Samples Bone Tissue Samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Adolescents: Individuals aged 10-19 years
- Young Adults: Individuals aged 20-39 years
- Elderly Adults: Individuals aged 40+ years

SUMMARY:
Guatemala has enforced mandatory fortification of sugar with vitamin A (VA) since June 1974 and has led to a highly successful reduction in VA deficiency and associated disease. However, Ribaya-Mercado et al. 2014, estimated the biological impact of sugar fortified with retinyl palmitate that there may be a risk of chronic excess intake of preformed VA associated with programs of mass fortification. A recent food consumption survey in two departments in Guatemala found the average daily sugar intake in children under the age of two who aren´t being breastfed is 30.3 g, which translates into a daily intake of 272 μg of retinol (almost the full estimated average requirement (EAR) for that age group). Since data from the second National Survey on Micronutrients suggest a risk of VA toxicity, it is important to determine the levels of hepatic VA directly in corpses of individuals, of all ages, who have died of non-metabolic causes. Due to this, the investigators propose to assess liver and bone VA levels in combination with gene expression, histopathology and biochemical analyses, to elicit indications of hypervitaminosis A in Guatemala.

DETAILED DESCRIPTION:
Objectives:

1. To determine the post mortem concentration of hepatic and bone VA in corpses of adolescent, young and elderly adults as an indicator of exposure to dietary VA
2. To assess the effect of high VA exposure on key enzymes in liver and bone tissue and to assess the risk of hypervitaminosis A in people exposed to compulsory mass vitamin A fortification program in Guatemala.

Methodology:

Setting and sampling The corpses for this study will be obtained from the National Institute of Forensic Sciences' (INACIF) departmental morgues in 2 hospitals in Guatemala City. The study population will be 150 cadavers sampled for VA tissue concentration; gene expression analysis combined with histopathology.

Sample collection process and duration All samples will be collected during necropsies carried out at the INACIF forensic morgue. During necropsy, the liver will be weighed and the information recorded. A range of up to 10 x 3 g samples of the liver's right lobe will be obtained. Each sample will be properly labelled with previously prepared codes. Liver samples for histopathological analysis will be stored in 10% buffered formalin for 24 hours prior to transfer to ethanol before embedding, sectioning and staining. All samples collected for retinoid analysis will be frozen on dry ice in the morgue, transported as such to the laboratory and subsequently stored at -80˚C. Liver samples for gene expression analysis will be collected in RNAlater solution to protect RNA stability and subsequently stored at -80˚C until shipment to Newcastle University. The hepatic VA analysis will be done in Newcastle University using established High Perfromance Liquid Chromatography (HPLC) methods. Samples for analysis of gene expression will be sent on dry ice to Newcastle for RNA extraction and quantification. Since it is possible to obtain good quality RNA suitable for Quantitative Polymerase Chain Reaction (q-PCR) based analyses from post mortem tissue up to 72 hours after death, tissue samples stored in RNAlater within 24 hours of death will be adequate for gene expression analysis. Furthermore, experience from the investigators human biobank in Newcastle shows that tissue RNA can be extracted successfully after the demise of a patient up to 72 hours after death as long as the tissue has a pH of over 6. Gene expression of key regulatory proteins, such as LRAT and CYP26A1 will be performed in Newcastle. Choice of genes was based on the fact that LRAT may become saturated at very high levels of VA, leading to increasing levels of free circulating VA that can be metabolized to retinoic acid and other metabolites via CYP26A. Histopathological analysis will be carried out by pathologists in Guatemala with digitised slides being sent to the pathologist within Newcastle University - these slides will be analysed by both pathologists independently.

Bone samples will also be obtained during the necropsy carried out at the INACIF forensic morgue. The iliac crest bone will be exposed by making an incision and removing the overlying soft tissue (skin, adipose tissue, connective tissue and muscle). The periosteum and cortical bone shall be removed via osteotomy exposing the spongy bone. Biopsy needles will be used to take samples from the spongy bone for analysis of tissue VA concentrations and gene expression, as previously described, at Newcastle University.

All samples will be shipped to Newcastle University on dry ice.

Study duration According to the information provided by INACIF 18 autopsies were performed between March and May 2013 on children less than one year of age, 24 on children from 1 to 4 years old, 11 on children 5 to 9 years old, 51 on individuals from 10 to 14 years old, 281 on adolescents 15 to 19 years old, and 401 on young adults 20 to 24 years old. According to INACIF's forensic doctor, ~60% of the total number of autopsies carried out in Guatemala are performed in the capital city. The main causes of death in children under the age of 9 were head injuries and other types of trauma. Individuals from 10 to 24 years of age died mainly due to violence: firearms, stabbings, choking and different types of trauma.

ELIGIBILITY:
Inclusion Criteria:

* Aged >10 years
* Non-metabolic cause of death (e.g. accidents, trauma, or violence from firearms, stabbings, cranial and other trauma, asphyxiation etc.)
* No longer than 24 hours since the time of death
* Lived in Guatemala (exposure to fortified sugar)

Exclusion Criteria:

* Aged <10 years
* Individuals with metabolic or nutritional conditions (diabetes, dyslipidemias, chronic alcoholism, etc.)
* Longer than 24 hours since the time of death
* Not Guatemalan resident (Tourist, visitor etc.)

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Guatemalan cadavers, from 2 hospitals in Guatemala City, aged >10 years with a non-metabolic cause of death, within 24 hours of death
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-10-24 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Liver Vitamin A concentration | Enrolment
  Liver Vitamin A concentration
Liver Gene Expression | Enrolment
  Gene expression associated with Vitamin A
Liver Histology | Enrolment
  Histological changes associated with Vitamin A
Bone Gene Expression | Enrolment
  Gene expression associated with Vitamin A

SECONDARY OUTCOMES:
Bone Vitamin A concentration | Enrolment
  Bone Vitamin A concentration

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Chew, MD, Principal Investigator — Institute of Nutrition of Central America and Panama; Erick Boy, MD, PhD, Principal Investigator — HarvestPlus; Georg Lietz, PhD, Study Director — Newcastle University
Locations (5):
- Guatemala (4):
  - Hospital Roosevelt, Guatemala City
  - INCAP, Guatemala City
  - Hospital General San Juan de Dios, Guatemala City
  - Morgue del INACIF, Guatemala City
- Newcastle University, Newcastle upon Tyne, Tyne and Wear, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pineda, O. (1998). Fortification of Sugar with Vitamin A. Food and Nutrition Bulletin, 19(2), 131-136.
- [Background] Ribaya-Mercado JD, Solomons NW, Medrano Y, Bulux J, Dolnikowski GG, Russell RM, Wallace CB. Use of the deuterated-retinol-dilution technique to monitor the vitamin A status of Nicaraguan schoolchildren 1 y after initiation of the Nicaraguan national program of sugar fortification with vitamin A. Am J Clin Nutr. 2004 Nov;80(5):1291-8. doi: 10.1093/ajcn/80.5.1291. PMID 15531678
- [Background] Olsen K, Suri DJ, Davis C, Sheftel J, Nishimoto K, Yamaoka Y, Toya Y, Welham NV, Tanumihardjo SA. Serum retinyl esters are positively correlated with analyzed total liver vitamin A reserves collected from US adults at time of death. Am J Clin Nutr. 2018 Nov 1;108(5):997-1005. doi: 10.1093/ajcn/nqy190. PMID 30475970